CLINICAL TRIAL: NCT04160897
Title: Risk of Hepatocellular Carcinoma in Patients Treated With ETV vs TDF for Chronic Hepatitis B With Compensated Cirrhosis: A Multicenter, Real-world and Respective Study
Brief Title: Risk of Hepatocellular Carcinoma in Patients Treated With ETV vs TDF for Chronic Hepatitis B With Compensated Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Qing XIe (Other)
Collaborators: Shanghai MedSci Healthcare Co. Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Qing XIe, Director of Department of Infectious Disease, Rui Jin Hospital, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: ISR-CN-9-10708
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis B, Chronic; Hepatocellular Carcinoma; Compensated Cirrhosis
Keywords: chronic hepatitis B; hepatocellular carcinoma; compensated cirrhosis; Chinese; entecavir; tenofovir disopropyl; multi-center; real-world; respective
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular | interventions — entecavir; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ETV cohort: CHB patients with entecavir naive treatment
  Interventions: Drug: Entecavir
- TDF cohort: CHB patients with naive tenofovir disopropyl naive treatment
  Interventions: Drug: Tenofovir Disoproxil

INTERVENTIONS:
Drug: Entecavir — entecavir naive for chronic hepatitis B patients
  Groups: ETV cohort
Drug: Tenofovir Disoproxil — tenofovir disopropyl naive for chronic hepatitis B patients
  Groups: TDF cohort

SUMMARY:
The current first-line treatment for HBV is long-term oral antiviral drugs to inhibit HBV DNA replication. First-line antiviral drugs recommended by the Chinese 2015 Hepatitis B Guidelines include ETV and TDF. This study is based on a real-world clinical cohort to retrospectively analyze the effects of ETV and TDF on the long-term (5-year) incidence of HCC in Chinese patients with chronic hepatitis B with compensated cirrhosis. The results will guide the revision of the Chinese HBV guidelines.

DETAILED DESCRIPTION:
HBV infection is a global problem, and China has a heavy disease burden with approximately 86 million people infected with HBV. According to the epidemiological survey of nearly 230,000 people in Northeast China in 2010-2013, the positive rate of HBsAg reached 6.1%, of which 10.7% had cirrhosis.

According to the latest authoritative guidelines, including the guidelines published in 2018 by American Association for the Study of Liver Diseases (AASLD) and in 2017 by European Association for the Study of Liver Diseases (EASL), entecavir (ETV) and tenofovir diisopropyl (TDF) are recommended as first-line antiviral drugs. ETV is a guanosine nucleoside analog that inhibits HBV polymerase and inhibits the synthesis of HBV DNA. TDF is a cyclic nucleoside phosphorylated diester structural analog of adenosine monophosphate, and its hydrolysis and phosphorylation products can inhibit the activity of HBV reverse transcriptase and also inhibit the synthesis of HBV DNA. In 2005, ETV was listed in China Mainland and TDF was listed in 2014. Over the years, clinical studies have shown that both have good antiviral effects and low drug resistance rates, so they are chosen as first-line antiviral drugs.

HBV infection is one of the risk factors for hepatocellular carcinoma (HCC). Previous studies based on the Chinese patients have shown that antiviral therapy (such as ETV) can significantly reduce the incidence of HCC in patients with cirrhosis (the 4-year cumulative incidence of HCC decreased from 17.5% to 9.4%). However, a study from South Korea published online in September 2018 in JAMA Oncology showed that TDF significantly reduced the incidence of HCC compared to ETV (HR 0.68, 95% CI 0.46-0.99) . In contrast, another multicenter study in Korea, published in March 2019 in The JOURNAL OF HEPATOLOGY showed no significant difference between ETV and TDF (HR 0.975, p=0.852) [4]. In the latter study, there was a problem with the small sample size, and the sample size was not sufficient to test the difference between the two antiviral drugs, and the sample size needed to be expanded to verify the result.

Compared with Koreans, the incidence of HCC in Chinese is significantly lower (in patients with cirrhosis, the 5-year cumulative incidence of HCC is about: China vs Korea: 12% vs 20%), showing the differences between countries. There is at present no similar study based on Chinese patients, especially in patients with cirrhosis to compare the effects of ETV and TDF on the incidence of HCC.

China has a huge disease burden and a high incidence of HCC. The ETV and TDF both have generic drugs marketing in China Mainland which through quality consistency evaluation and entering the 4+7 drug procurement (the centralized drug procurement in "4+7 Cities": Beijing, Tianjin, Shanghai, Chongqing, Shenyang, Dalian, Xiamen, Guangzhou, Shenzhen, Chengdu and Xian), bringing good antiviral effect to patients at preferential prices. If we can detect the difference in the occurrence of HCC between ETV and TDF, rational selection of drugs will reduce the incidence of HCC in Chinese patients with chronic hepatitis B (Korean studies showed that cumulative HCC patients can reduce 32% in 5 years), greatly reducing the burden on Chinese patients and health care.

This research is a real-world, multi-center, retrospective, and observational study.

Patient data are collected from 5-10 research centers in mainland China, including basic demographic information, antiviral regimen, time of stating antivirus, endpoint event, time of endpoint event, last follow-up time, important testing data, etc.

Patients with the time of last follow-up (or the time of the endpoint event) between 2013-1-1 and 2019-12-31 are included in this study.

Based on the data we collect, the Propensity Score Matching and Inverse Probability Multiple Weighted methods and the Competing Risk Model are utilized to correct the confounding factors to calculate the impact of TDF and ETV on HCC events.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg+ > 6 months
* age 18-80
* TDF or ETV Treatment Naive
* cirrhosis

Exclusion Criteria:

* TDF/ETV treatment duration<12 m
* decompensated cirrhosis
* previous H/O organ or stem cell transplant
* IFN exposure or combination of IFN>4 w
* HCC, death or OLT within 12 m after TDF or ETV treatment;
* previous HCC history;
* key data (such as key medical history, hematological and biochemical tests, HBV DNA and HBV antibody/antigen before treatment, et al) missing or error.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted in high-risk populations of HCC (patients with cirrhosis). According to the studies from Taiwan and Hongkong, the cumulative incidence of HCC in Chinese patients with cirrhosis in the ETV group was about 11.8-13.8% over 5 years, and we estimate it to be 12.8%; the 5-year incidence of HCC in the TDF group is estimated to be 8.0% according to the studies from Korea with the HR=0.55-0.75. Actual patients' use of ETV and TDF in China is about 3:1. We calculated that for this study to have 80% power to detect a 5% relative difference between the TDF and ETV groups, there would have to be 202 events and enroll 539 and 1616 patients at least in TDF and ETV treatment group based on log-rank (Lakatos) test.
  On the basis of these calculations, we planned to enroll 4,000 patients (1,000 patients in the TDF group, 3,000 patients in the ETV group).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
The 5-year cumulative incidence of hepatocellular carcinoma | 5 years
  Compare the difference in the 5-year cumulative incidence of HCC in Chinese patients with chronic hepatitis B with cirrhosis in real world between ETV and TDF.

SECONDARY OUTCOMES:
The 5-year cumulative all-cause mortality rate | 5 years
  Compare the difference in the 5-year cumulative all-cause mortality rate in Chinese patients with chronic hepatitis B with cirrhosis in real world between ETV and TDF.
The 5-year cumulative liver transplantation rate | 5 years
  Compare the difference in the 5-year cumulative liver transplantation rate in Chinese patients with chronic hepatitis B with cirrhosis in real world between ETV and TDF.
The 5-year cumulative liver disease-related mortality | 5 years
  Compare the difference in the 5-year cumulative liver disease-related mortality in Chinese patients with chronic hepatitis B with cirrhosis in real world between ETV and TDF.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xie, MD, Study Chair — Director of Department of Infectious Disease, Rui Jin Hospital
Locations (1):
- Rui Jin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Q, Qi W, Wang X, Zhang Y, Xu Y, Qin S, Zhao P, Guo H, Jiao J, Zhou C, Ji S, Wang J. Epidemiology of Hepatitis B and Hepatitis C Infections and Benefits of Programs for Hepatitis Prevention in Northeastern China: A Cross-Sectional Study. Clin Infect Dis. 2016 Feb 1;62(3):305-12. doi: 10.1093/cid/civ859. Epub 2015 Oct 3. PMID 26433720
- [Background] Su TH, Hu TH, Chen CY, Huang YH, Chuang WL, Lin CC, Wang CC, Su WW, Chen MY, Peng CY, Chien RN, Huang YW, Wang HY, Lin CL, Yang SS, Chen TM, Mo LR, Hsu SJ, Tseng KC, Hsieh TY, Suk FM, Hu CT, Bair MJ, Liang CC, Lei YC, Tseng TC, Chen CL, Kao JH; C-TEAM study group and the Taiwan Liver Diseases Consortium. Four-year entecavir therapy reduces hepatocellular carcinoma, cirrhotic events and mortality in chronic hepatitis B patients. Liver Int. 2016 Dec;36(12):1755-1764. doi: 10.1111/liv.13253. Epub 2016 Oct 4. PMID 27634134
- [Background] Choi J, Kim HJ, Lee J, Cho S, Ko MJ, Lim YS. Risk of Hepatocellular Carcinoma in Patients Treated With Entecavir vs Tenofovir for Chronic Hepatitis B: A Korean Nationwide Cohort Study. JAMA Oncol. 2019 Jan 1;5(1):30-36. doi: 10.1001/jamaoncol.2018.4070. PMID 30267080
- [Background] Kim SU, Seo YS, Lee HA, Kim MN, Lee YR, Lee HW, Park JY, Kim DY, Ahn SH, Han KH, Hwang SG, Rim KS, Um SH, Tak WY, Kweon YO, Kim BK, Park SY. A multicenter study of entecavir vs. tenofovir on prognosis of treatment-naive chronic hepatitis B in South Korea. J Hepatol. 2019 Sep;71(3):456-464. doi: 10.1016/j.jhep.2019.03.028. Epub 2019 Apr 6. PMID 30959156
- [Background] Wong GL, Chan HL, Mak CW, Lee SK, Ip ZM, Lam AT, Iu HW, Leung JM, Lai JW, Lo AO, Chan HY, Wong VW. Entecavir treatment reduces hepatic events and deaths in chronic hepatitis B patients with liver cirrhosis. Hepatology. 2013 Nov;58(5):1537-47. doi: 10.1002/hep.26301. Epub 2013 Sep 30. PMID 23389810
- [Background] Chinese Society of Hepatology, Chinese Medical Association; Chinese Society of Infectious Diseases, Chinese Medical Association; Hou JL, lai W. [The guideline of prevention and treatment for chronic hepatitis B: a 2015 update]. Zhonghua Gan Zang Bing Za Zhi. 2015 Dec;23(12):888-905. doi: 10.3760/cma.j.issn.1007-3418.2015.12.002. No abstract available. Chinese. PMID 26739464
- [Background] Chinese Foundation for Hepatitis Prevention and Control; Chinese Society of Infectious Disease and Chinese Society of Hepatology, Chinese Medical Association; Liver Disease Committee of Chinese Research Hospital Association. [Consensus on clinical application of transient elastography detecting liver fibrosis: a 2018 update]. Zhonghua Gan Zang Bing Za Zhi. 2019 Mar 20;27(3):182-191. doi: 10.3760/cma.j.issn.1007-3418.2019.03.004. Chinese. PMID 30929334